CLINICAL TRIAL: NCT03418701
Title: Culturally Sensitive Primary Care Clinic-based Interventions by Community Health Workers and Trained Physicians to Promote and Sustain Weight Loss Among Obese Black Women Patients
Brief Title: Health-Smart for Weight Loss at UF Jax Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201703386; AD-1609-36187 (Other Grant/Funding Number: PATIENT-CENTERED OUTCOMES RES INST)
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: Women's health
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Centered Culturally Sensitive WLM (Active Comparator): This program is designed to enable physicians to: (a) talk with their patients about their weight, weight loss goals, goal barriers, strategies for overcoming these barriers, and deliver this talk in patient-centered, culturally sensitive ways, (b) assist their patients with engaging in self-identified strategies for achieving and sustaining their self selected goals for weight loss and overall health, (c) be knowledgeable about health-smart behaviors, (d) use behaviors and display attitudes in physician-patient interactions with patients that are provider cultural sensitivity indicators in published literature, and (e) say and display behaviors and attitudes that patients identified as important when discussing obesity and losing weight.
  Interventions: Behavioral: Health Smart for Weight Loss
- Standard Behavioral WLM (Active Comparator): This program is designed to enable physicians to: (a) implement motivational interviewing approaches when talking with their patients about their weight loss goals and behavioral strategies to achieve these goals, (b) become knowledgeable about empirically supported behavioral change principles that have been used to help patients maintain weight loss in previous interventions, (c) communicate how to use these empirically supported behavioral change principles to have patients initiate or maintain their self-selected health-smart goals related to weight loss and/or weight loss maintenance, and (d) use motivational interviewing approaches to communicate empathy and understanding with patients who are struggling to maintain their weight loss and/or accomplish a behavioral goal.
  Interventions: Behavioral: Health Smart for Weight Loss

INTERVENTIONS:
Behavioral: Health Smart for Weight Loss — We will test the effectiveness of a culturally sensitive, evidence-based, multi-component, behavioral program for treating obesity called Health-Smart. This program will be implemented for 6 months in 20 UF Health Jacksonville primary care clinics by Community Health Workers (CHWs) with Black women patients who have obesity, and followed by either of two physician-implemented behavioral counseling weight loss maintenance programs that are applied quarterly over 12 months to prevent weight gain. Specifically, we will compare the effects on weight-loss and weight-loss maintenance of (1) Health-Smart plus the Patient-Centered, Culturally Sensitive Weight Loss Maintenance Program (PCS-WLM), and (2) Health-Smart plus the Standard Behavioral Weight Loss Maintenance Program (SB-WLM).

SUMMARY:
The study will test the effectiveness of a culturally sensitive, evidence-based, multi-component, behavioral program for treating obesity called Health-Smart. This program is being implemented by Community Health Workers at the primary care centers and followed by either of two physician-implemented behavioral counseling programs to prevent weight gain--programs that are implemented quarterly over 12 months.

DETAILED DESCRIPTION:
Objectives: Aim 1 was to evaluate the effectiveness of the community health worker (CHW)-implemented, clinic-located, evidence-based, 6-month Health-Smart Weight Loss (HSWL) Program, as indicated by participants' mean weight loss. Aim 2 was to compare the outcomes of the following two 12-month, clinic-based weight loss maintenance programs implemented by patients' physicians after these patients completed the 6-month weight loss intervention: the physician-implemented Patient-Centered, Culturally Sensitive Weight Loss Maintenance (PCCS-WLM) intervention, and the Standard Behavioral Weight Loss Maintenance (SB-WLM) intervention. These two weight loss maintenance interventions differ in that the physicians who implemented the PCCS-WLM intervention were trained to display patient-identified, culturally sensitive behaviors and attitudes when talking with patients about their weight and to support patients' engagement in health promoting (health-smart) behaviors in order to promote patients' weight loss maintenance, whereas physicians in the SB-WLM intervention were trained to use behavioral change principles and skills as well as motivational interviewing approaches to behavior change in order to promote patients' weight loss maintenance. Aim 3 was to implement and evaluate a medical assistant-led program to integrate CHWs into health care teams.

Methods: Participants were recruited from 21 primary care practices operated by an academic medical center. Participants' eligibility criteria were: Black women ages 21 years or older with a BMI of 30 kg/m2 or higher who had at least 2 clinic visits in the previous 24 months and were ready to change their diet and physical activity level.

All participants received the 6-month CHW-implemented HSWL Program to address Aim 1. Therefore, results from baseline to 6 months are presented as one group. The study was constructed as a cluster-randomized trial to address Aim 2; thus, after the HSWL Program involving all participants was completed, clinics were randomized to the either the SB-WLM group or the PCCS-WLM group. Consequently, results after 6 months are presented separately for the two groups. Clinics were randomized with patients nested within clinic.

To address Aim 1, a paired samples t-test and confidence interval of the proportion of the sample that achieved 5% or more weight loss by 6 months were used. To address Aim 2, a logistic regression with participants nested within clinics and Aim 2 study group as the independent variable was used. To address Aim 3, which was to evaluate integration of CHWs into the health care team, a virtual meeting was held with the CHWs who remained at the end of the study (n=8) for the purpose of asking exploratory semi-structured questions about the clinical staff behaviors that helped them feel or not feel integrated into the clinical team and to identify what would improve and/or sustain integration of CHWs into the clinical team. Content analysis using the constant comparison method was applied to the responses of the CHWs to the semi-structured questions asked. The communications and follow-through subscale of the TeamSTEPPS Assessment Tool was used to assess communication among the clinic staff as viewed by the participating clinic staff as a group and CHWs as a group. Mean ratings of responses to this subscale for each of these groups were calculated.

ELIGIBILITY:
Inclusion Criteria:

* African American/black
* Female
* Age 21 years or older
* BMI range ≥ 30kg/m2 (5) active patient of a participating clinic (i.e., at least 2 clinic visits in the last 24 months)
* Willing and ready to change one's diet and physical activity level
* Willing to be randomized to either of the two weight-loss maintenance intervention groups

Exclusion Criteria:

* Any serious medical condition that likely affects weight, such as end stage renal disease or cancer
* Prior bariatric surgery within the last 5 years or plans for this surgery in the next 2 years
* Use of prescription or over-the-counter weight-loss medication within the last 6 months
* Pregnant or plan to get pregnant within the next 2 years
* Plan to relocate from the area within the next 2 years
* Having had unintentional weight loss (>or = to 5% of body weight) within 6 months prior to enrollment
* Taking a daily dose of oral corticosteroid antipsychotic (clozapine, olanzapine, or risperidone) for less than 6 months

Ages: 21 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Tucker, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health Jacksonville Primary Care network, Jacksonville, Florida, United States

REFERENCES:
- [Result] Tucker CM, Anton SD, Wippold GM, Marsiske M, Bilello LA, Henry MA, Shah NR, Gautam SP, Klein KG, Mathews A, Webb F, Desmond F. Promoting weight-loss maintenance among Black women primary care patients: A cluster RCT of a culturally sensitive versus standard behavioural approach. Clin Obes. 2022 Dec;12(6):e12553. doi: 10.1111/cob.12553. Epub 2022 Sep 23. PMID 36151609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multifaceted approach was used to recruit Black women patients with obesity from the participating primary care centers. Recruitment included distribution of marketing materials in the clinic waiting rooms and exam rooms. Providers also discussed the trial with potentially eligible patients if they had an appointment during the recruitment period. If a patient showed interest in participating, she was to complete a form allowing a study team member to contact her about the trial.
Pre-assignment Details: A research coordinator performed a screening interview after receiving verbal consent from the caller. If the caller met the screening criteria and wants to participate in the study, a visit with their physician was scheduled to ensure that there were no medical contraindications to participation. This screening visit included a review of the patient's medications, medical history and physical exam. At the end of the screening visit, patients were informed whether they qualified for the study.
Units Other Than Participants: clinics
Groups:
- Phase 1: 6-month CHW-implemented HSWL Program: All participants started in the HSWL program where they went to CHW led sessions that occurred weekly for 3 months then biweekly for 3 months. . During these sessions, the participants viewed and discussed segments of an HSWL Program DVD that shows culturally diverse families and community members, physicians, and other health care providers discussing health-smart behaviors and real-world strategies for engaging in these behaviors. The participants were given an HSWL Program Resource Guide, which is a supplement to the DVD, that contains more detailed information about the discussed health-smart behaviors. These participants were asked to read short sections of this guide to prepare them for the next group discussion. An important aspect of the group sessions was that participants learned from and taught each other ways to consistently engage in health-smart behaviors, including ways to overcome barriers to these behaviors. The CHWs facilitated these discussions called attention to relevant information in the DVD and resource guide only when needed.
- Phase 2: Patient Centered Culturally Sensitive WLM: This program is designed to enable physicians to: (a) talk with their patients about their weight, weight loss goals, goal barriers, strategies for overcoming barriers, and talk in patient-centered, culturally sensitive ways, (b) assist patients with engaging in self-identified strategies for achieving and sustaining their goals for weight loss and overall health, (c) be knowledgeable about health-smart behaviors, (d) use behaviors and display attitudes in physician-patient interactions that are provider cultural sensitivity indicators and (e) say and display behaviors/attitudes that patients identified as important when discussing obesity and losing weight.
  Health Smart for Weight Loss: We will test the effectiveness of a culturally sensitive, evidence-based, multi-component, behavioral program for treating obesity called Health-Smart. This program will be implemented for 6 months in 20 UF Health Jacksonville primary care clinics by Community Health Workers (CHWs) with Black women patients who have obesity, and followed by either of two physician-implemented behavioral counseling weight loss maintenance programs that are applied quarterly over 12 months to prevent weight gain. Specifically, we will compare the effects on weight-loss and weight-loss maintenance of (1) Health-Smart plus the Patient-Centered, Culturally Sensitive Weight Loss Maintenance Program (PCS-WLM), and (2) Health-Smart plus the Standard Behavioral Weight Loss Maintenance Program (SB-WLM).
- Phase 2:Standard Behavioral WLM: This program is designed to enable physicians to: (a) implement motivational interviewing approaches with their patients about their weight loss goals and behavioral strategies to achieve these goals, (b) become knowledgeable about behavioral change principles that have been used to help patients maintain weight loss, (c) communicate how to use these behavioral change principles to have patients initiate or maintain their health-smart goals related to weight loss and/or weight loss maintenance, and (d) use motivational interviewing approaches to communicate empathy with patients who are struggling to maintain their weight loss and/or accomplish a behavioral goal.
  Health Smart for Weight Loss: We will test the effectiveness of a culturally sensitive, evidence-based, multi-component, behavioral program for treating obesity called Health-Smart. This program will be implemented for 6 months in 20 UF Health Jacksonville primary care clinics by Community Health Workers (CHWs) with Black women patients who have obesity, and followed by either of two physician-implemented behavioral counseling weight loss maintenance programs that are applied quarterly over 12 months to prevent weight gain. Specifically, we will compare the effects on weight-loss and weight-loss maintenance of (1) Health-Smart plus the Patient-Centered, Culturally Sensitive Weight Loss Maintenance Program (PCS-WLM), and (2) Health-Smart plus the Standard Behavioral Weight Loss Maintenance Program (SB-WLM).
Period: Phase 1: 6-mo CHW-implemented HSWL Progr
Arm/Group | Phase 1: 6-month CHW-implemented HSWL Program | Phase 2: Patient Centered Culturally Sensitive WLM | Phase 2:Standard Behavioral WLM
Started | 683; 20 clinics | 0; 0 clinics | 0; 0 clinics
Completed | 356; 20 clinics | 0; 0 clinics | 0; 0 clinics
Not Completed | 327; 0 clinics | 0; 0 clinics | 0; 0 clinics
Period: Phase 2: 12-mo Weight Loss Maintenance
Arm/Group | Phase 1: 6-month CHW-implemented HSWL Program | Phase 2: Patient Centered Culturally Sensitive WLM | Phase 2:Standard Behavioral WLM
Started | 0; 0 clinics | 183; 10 clinics | 173; 10 clinics
Completed | 0; 0 clinics | 140; 10 clinics | 131; 10 clinics
Not Completed | 0; 0 clinics | 43; 0 clinics | 42; 0 clinics

BASELINE CHARACTERISTICS:
Population: All participants were black women patients from participating primary care centers
Groups:
- Patient Centered Culturally Sensitive WLM: This program is designed to enable physicians to: (a) talk with their patients about their weight, weight loss goals, goal barriers, strategies for overcoming barriers, and talk in patient-centered, culturally sensitive ways, (b) assist patients with engaging in self-identified strategies for achieving and sustaining their goals for weight loss and overall health, (c) be knowledgeable about health-smart behaviors, (d) use behaviors and display attitudes in physician-patient interactions that are provider cultural sensitivity indicators and (e) say and display behaviors/attitudes that patients identified as important when discussing obesity and losing weight.
  Health Smart for Weight Loss: We will test the effectiveness of a culturally sensitive, evidence-based, multi-component, behavioral program for treating obesity called Health-Smart. This program will be implemented for 6 months in 20 UF Health Jacksonville primary care clinics by Community Health Workers (CHWs) with Black women patients who have obesity, and followed by either of two physician-implemented behavioral counseling weight loss maintenance programs that are applied quarterly over 12 months to prevent weight gain. Specifically, we will compare the effects on weight-loss and weight-loss maintenance of (1) Health-Smart plus the Patient-Centered, Culturally Sensitive Weight Loss Maintenance Program (PCS-WLM), and (2) Health-Smart plus the Standard Behavioral Weight Loss Maintenance Program (SB-WLM).
- Standard Behavioral WLM: This program is designed to enable physicians to: (a) implement motivational interviewing approaches with their patients about their weight loss goals and behavioral strategies to achieve these goals, (b) become knowledgeable about behavioral change principles that have been used to help patients maintain weight loss, (c) communicate how to use these behavioral change principles to have patients initiate or maintain their health-smart goals related to weight loss and/or weight loss maintenance, and (d) use motivational interviewing approaches to communicate empathy with patients who are struggling to maintain their weight loss and/or accomplish a behavioral goal.
  Health Smart for Weight Loss: We will test the effectiveness of a culturally sensitive, evidence-based, multi-component, behavioral program for treating obesity called Health-Smart. This program will be implemented for 6 months in 20 UF Health Jacksonville primary care clinics by Community Health Workers (CHWs) with Black women patients who have obesity, and followed by either of two physician-implemented behavioral counseling weight loss maintenance programs that are applied quarterly over 12 months to prevent weight gain. Specifically, we will compare the effects on weight-loss and weight-loss maintenance of (1) Health-Smart plus the Patient-Centered, Culturally Sensitive Weight Loss Maintenance Program (PCS-WLM), and (2) Health-Smart plus the Standard Behavioral Weight Loss Maintenance Program (SB-WLM).
- Total: Total of all reporting groups
Arm/Group | Patient Centered Culturally Sensitive WLM | Standard Behavioral WLM | Total
Number analyzed (Participants) | 351 | 332 | 683
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.46 (12.32) | 51.52 (12.06) | 52.04 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 351 | 332 | 683
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 351 | 332 | 683
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 351 | 332 | 683
Weight [Mean (Standard Deviation); unit: pounds] | 235.8 (47.8) | 242.3 (52.1) | 240 (51.7)

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: percentage of participating patients who show clinically significant weight loss (i.e., at least 5% of baseline body weight)
Time Frame: 6 months
Population: In order to determine the significance of the proportion of participants who achieved 5% weight loss from baseline to 6 months, a confidence interval of the proportion was used. A dichotomized dependent variable was used where 0 indicated that the participant did not achieve 5% or more weight loss and 1 indicated that the participant achieved 5% or more. No covariates were used.
Measure: Number (95% Confidence Interval); unit: percent who lost 5% or more weight
Groups:
- 6-month CHW-implemented HSWL Program: This program is designed to enable physicians to: (a) talk with their patients about their weight, weight loss goals, goal barriers, strategies for overcoming barriers, and talk in patient-centered, culturally sensitive ways, (b) assist patients with engaging in self-identified strategies for achieving and sustaining their goals for weight loss and overall health, (c) be knowledgeable about health-smart behaviors, (d) use behaviors and display attitudes in physician-patient interactions that are provider cultural sensitivity indicators and (e) say and display behaviors/attitudes that patients identified as important when discussing obesity and losing weight.
  Health Smart for Weight Loss: We will test the effectiveness of a culturally sensitive, evidence-based, multi-component, behavioral program for treating obesity called Health-Smart. This program will be implemented for 6 months in 20 UF Health Jacksonville primary care clinics by Community Health Workers (CHWs) with Black women patients who have obesity, and followed by either of two physician-implemented behavioral counseling weight loss maintenance programs that are applied quarterly over 12 months to prevent weight gain. Specifically, we will compare the effects on weight-loss and weight-loss maintenance of (1) Health-Smart plus the Patient-Centered, Culturally Sensitive Weight Loss Maintenance Program (PCS-WLM), and (2) Health-Smart plus the Standard Behavioral Weight Loss Maintenance Program (SB-WLM).
Arm/Group | 6-month CHW-implemented HSWL Program
Number analyzed (Participants) | 356
percent who lost 5% or more weight | 24.04 [19.3 to 29.4]
Statistical Analysis 1: Comparison: 6-month CHW-implemented HSWL Program; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 2.67, 95% CI 2-sided [0.93 to 4.40]

2. Primary Outcome: Weight Loss Maintenance
Description: percentage of participants will maintain initial weight loss or show continued weight loss
Time Frame: 18 months
Population: Main analysis was a multilevel logistic regression with participants nested within clinic. A dichotomized dependent variable was used where 0 indicated that the participant gained more than 1 pound between 6 and 18 months (i.e., did not maintain weight loss) and 1 indicated that the participant gained less than 1 pound or continued to lose weight between 6 and 18 months (i.e., maintained weight loss). The independent variable was weight loss maintenance group. No covariates were used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patient Centered Culturally Sensitive WLM | Standard Behavioral WLM
Number analyzed (Participants) | 140 | 131
percentage of participants | 34.63 [25.8 to 44.2] | 29.48 [21.9 to 37.5]
Statistical Analysis 1: Comparison: Patient Centered Culturally Sensitive WLM vs Standard Behavioral WLM; Test type: Superiority; p < 0.05, Mixed Models Analysis; A multilevel logistic regression with participants nested within clinic; Odds Ratio, log = 0.47, 95% CI 2-sided [0.22 to 1.15]

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events were reported to the community health workers during the Health-Smart weekly sessions in Phase 1 and then to physicians in Phase 2. Adverse events were considered serious if they resulted in hospitalizations.
Groups:
- 6-month CHW-implemented HSWL Program: All participants started in the HSWL program where they went to CHW led sessions that occurred weekly for 3 months then biweekly for 3 months. . During these sessions, the participants viewed and discussed segments of an HSWL Program DVD that shows culturally diverse families and community members, physicians, and other health care providers discussing health-smart behaviors and real-world strategies for engaging in these behaviors. The participants were given an HSWL Program Resource Guide, which is a supplement to the DVD, that contains more detailed information about the discussed health-smart behaviors. These participants were asked to read short sections of this guide to prepare them for the next group discussion. An important aspect of the group sessions was that participants learned from and taught each other ways to consistently engage in health-smart behaviors, including ways to overcome barriers to these behaviors. The CHWs facilitated these discussions called attention to relevant information in the DVD and resource guide only when needed.
Arm/Group | 6-month CHW-implemented HSWL Program | Patient Centered Culturally Sensitive WLM | Standard Behavioral WLM
All-Cause Mortality (participants affected / at risk) | 1/683 | 2/183 | 2/173
Serious Adverse Events (participants affected / at risk) | 5/683 | 0/183 | 0/173
Other Adverse Events (participants affected / at risk) | 3/683 | 0/183 | 0/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6-month CHW-implemented HSWL Program (N=683) | Patient Centered Culturally Sensitive WLM (N=183) | Standard Behavioral WLM (N=173)
back surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
knee arthroplasty (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
nephrostolithotomy surgery (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6-month CHW-implemented HSWL Program (N=683) | Patient Centered Culturally Sensitive WLM (N=183) | Standard Behavioral WLM (N=173)
motor vehicle accident with minor injuries (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fell in store parking lot (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
cyst drainage (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Since the intervention delivered as part of Aim 1 was an uncontrolled pre-post study, we cannot determine whether or not the HSWL intervention caused the weight loss observed among our study participants during the first six months, as there was not a control/comparison group.

Another limitation is that of the 683 Black women who enrolled and provided baseline data, only 63.9% actually participated in the study intervention (i.e., attended any of the interventions sessions in the study).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT03418701/Prot_SAP_000.pdf